CLINICAL TRIAL: NCT05866276
Title: A Real-World Multicentre Prospective Study to Determine the Accuracy of the SCORED (SCreening for Occult REnal Disease) Questionnaire for SCreening REnal Risk Early Against Nephropathy in Adult Population in Asia
Brief Title: To Determine the Accuracy of SCreening for Occult REnal Disease (SCORED) Questionnaire for CKD Risk Among Asian Patients
Acronym: SCREEN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00353
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the accuracy of SCreening for Occult REnal Disease (SCORED) questionnaire for CKD risk among Asian Patients

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Normal Adult Population in Asia
Sampling Method: Non-Probability Sample
Enrollment: 1426 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 28 February 2024
  The primary objective is to evaluate the accuracy of SCORED tool in identifying individuals at risk for the development of CKD in the Asian population. The primary outcomes, sensitivity, and specificity will be summarised using percentage and 95% confidence intervals to be measured at Baseline up to 6months after enrollment

CONTACTS AND LOCATIONS:
Locations (3):
- Indonesia (2):
  - Perisai Husada, Bandung, West Java
  - Research Site, Surabaya
- Nguyen Tri Phuong Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- See also: D1843R00353_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00353&attachmentIdentifier=e5cd71e7-cd83-40b1-b571-0bdb071671f0&fileName=D1843R00353_CSR_Synopsis_Redacted.pdf&versionIdentifier=